CLINICAL TRIAL: NCT02604303
Title: A Prospective Analysis on the Expansion Rates of Abdominal Aortic Aneurysms
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: VA Northern California Health Care System (U.S. Federal Agency)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Other Study IDs: Medtronic A1231656
Record Dates: First submitted 2015-10-06; First posted 2015-11-13 (Estimated); Last update posted 2019-11-29 (Actual); Status verified 2019-11

CONDITIONS: Abdominal Aortic Aneurysm
Keywords: Abdominal Aortic Aneurysm; RhoA; Biomarker
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Patient monocytes from peripheral blood
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: No Intervention — No intervention; prospective observational study

SUMMARY:
Abdominal aortic aneurysm (AAA) disease is an abnormal bulging of the main abdominal artery, which is the called the abdominal aorta. The purpose of this observational study is to identify whether a blood biomarker protein RhoA can predict which small AAA patients may need surgery in the future.

Participating patients will receive an ultrasound and blood draw. The patients will be divided into expanding and stable aorta groups after determining each patient's aortic expansion rate. The blood RhoA levels and aortic expansion rates between both groups would then be compared to look for any relationships.

DETAILED DESCRIPTION:
Abdominal aortic aneurysm (AAA) is an asymptomatic problem until rupture occurs, causing excruciating pain and sudden death. It is diagnosed typically by ultrasound when the aortic diameter is ≥ 3.0 cm and an aortic diameter ≥ 5.5 cm generally requires surgical repair to prevent rupture. A normal aorta is 2.0 cm in diameter. For patients with small AAA (3.0-5.4 cm) serial imaging studies is recommended along with risk factor modification. However, follow up ultrasound protocols are difficult to follow, resulting in many patients with expanding AAA not being detected until too late. To streamline and better identify patients with small AAAs at risk for expansion, the investigators look to RhoA as a possible biomarker.

The investigators will recruit within a 3-year period a total of 200 subjects diagnosed with small AAA 3.0-5.4 cm diameter from the VA Northern California Health Care System. All subjects enrolled will already have a baseline aortic diameter established at the time of initial AAA screening or diagnostic imaging. The investigators expect the follow up ultrasound measurement for this study will be at least 1 to 5 years after their baseline ultrasound study. The follow up evaluation will then assess expansion rates of the aorta. Stable aorta subjects will have an expansion rate of less than 0.2 cm/year and expanding aorta subjects will have an expansion rate ≥ 0.2 cm/year as based on preliminary data. After the ultrasound, 30 ml of blood will be drawn into heparinized tubes and undergo blood analysis for the RhoA protein in monocytes. All patients will be notified of the possible need to return back for either clinical reason: AAA greater than 5.5 cm or research protocol reasons: inadequate monocyte collection or changing clinical data requirements. Cardiovascular risk factors will also be collected. All collected data between stable and expanding AAA groups will then be compared for analysis.

If biological or clinical risk factors are identified as reliable biomarkers for AAA expansion, then AAA screening programs could be modified to increase screening yield and improve surveillance for small AAAs. Additionally, novel diagnostic techniques could be developed to better identify small AAA patients at risk for surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Over the age of 21 years.
2. Have been screened for abdominal aortic aneurysm by the VA or found to have an aorta visualized from diagnostic imaging at least once.
3. Currently on no medications which would interfere with wound healing or compromise the blood draw.
4. Not pregnant nor planning to become pregnant during study period.
5. No previous history of AAA repair.

Exclusion Criteria:

1. Failure to meet inclusion criteria.
2. Patient withdraws from the study.
3. In the opinion of the principle investigator, multiple comorbidities that make analysis difficult.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Veterans of VA Northern California Health Care System
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2015-09; Primary Completion 2020-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Aortic Expansion Rate | Immediately after study ultrasound for each subject. The aortic expansion rate is immediately obtained once the study ultrasound measurement of the aortic diameter is verified.
  Aortic expansion rate (cm/yr) is calculated by taking the difference of aortic growth (cm) divided by the number of days between a patient's screening date and the study date. This rate is then converted into cm/yr.

SECONDARY OUTCOMES:
RhoA levels | From collection of blood to completion of blood analysis. This analysis takes 5-7 days to complete per patient.
  RhoA levels measured in fluorescent units from patient monocytes will be determined

CONTACTS AND LOCATIONS:
Overall Officials: Eugene S Lee, MD, PhD, Principal Investigator — VA Northern California Health Care System
Locations (1):
- Sacramento VA Medical Center, Mather, California, United States